CLINICAL TRIAL: NCT06077435
Title: Comparative Analysis of AI Software and Conventional Colonoscopy for Enhanced Polyp Detection and Diagnosis: A Randomized Controlled Trial
Brief Title: Comparative Analysis of AI Software for Enhanced Polyp Detection and Diagnosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Jonas Varkey, Principal investigator, Senior Consultant, MD, PhD,, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 981840
Record Dates: First submitted 2023-09-27; First posted 2023-10-11 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Colonic Polyp; Colon Lesion
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CAD-EYE (Active Comparator): AI system 1. Sealed envelopes in blocks of four were used for randomisation.
  Interventions: Device: AI
- GI-GENIUS (Active Comparator): AI system 2. Sealed envelopes in blocks of four were used for randomisation
  Interventions: Device: AI
- Endo-AID (Active Comparator): AI system 3. Sealed envelopes in blocks of four were used for randomisation
  Interventions: Device: AI
- No AI (No Intervention): No AI. conventional examination. Sealed envelopes in blocks of four were used for randomisation

INTERVENTIONS:
Device: AI — AI system
  Arms: CAD-EYE; Endo-AID; GI-GENIUS

SUMMARY:
Purpose & Research Questions

The purpose of this study is to evaluate whether artificial intelligence (AI) improves the detection of polyps and whether the system can classify the type and severity of detected changes. The investigators will also assess if there are any differences between the various AI systems and whether the polyps that may be missed are benign or malignant.

DETAILED DESCRIPTION:
Materials: Selection, Representativeness, and Grouping

The study is a randomized controlled clinical trial conducted at Västra Götaland region. Patients are randomized to receive either AI or conventional endoscopy, and each endoscopy unit has access to at least one AI device. Informed consent is obtained from patients before the examination.

Before the examination, patients are asked if they want to participate in the study. If the patient wishes to participate, informed consent is obtained. The endoscopist then draws a slip from an envelope, determining whether conventional colonoscopy or AI will be used. During conventional colonoscopy, the patient is examined according to routine practice. After the examination, a questionnaire is filled out, recording various findings from the examination. During AI examinations, the AI system is activated only during instrument withdrawal. The system identifies polyps and alerts the endoscopist. Additionally, two of the AI systems (GI-Genius, CADEYE) have the ability to characterize the detected polyps and provide an interpretation of whether the changes are benign or malignant. After the examination, a similar questionnaire is completed as in conventional colonoscopy.

Method: Data Collection

Basic data will be recorded, including the reason for the examination, other illnesses, medications, demographic data such as gender, age, family history of cancer, and the time of the examination (morning or afternoon). During the examination, the following will be recorded: the number of polyps, macroscopic classification of polyps, AI system's characterization of the polyps, bowel cleansing quality, laxative method, medication during the examination, complications occurring during or after the examination. Withdrawal time is recorded, as well as the number of false-positive polyps and supplementation with histological data of polyps after review by the pathologist. All materials and costs associated with the examination are recorded.

Three different AI systems will be used at the various hospital sites, namely EndoAid (Olympus), CADEYE (Fujinon), and GI-Genius (Medtronic). All units will randomize each examination to either AI or non-AI.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Elective colonoscopy

Exclusion Criteria:

* Patient declines to participate in the study.
* Age < 50 years
* Unprepared bowel

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 915 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
To compare the effectiveness of AI systems in characterizing polyps with conventional histology | During procedure (5minutes)
  The endoscopist's ability to characterize lesions with and without AI will be assessed, and this assessment will be compared to histology
Comparison of Adenoma Detection Rates (ADR) between colonoscopies assisted by Artificial Intelligence (AI) and conventional colonoscopies without AI | During procedure (up to 40 minutes)
  The ADR is typically expressed as a percentage and is calculated using the following formula:Number of colonoscopies with adenoma detection/ Total number of colonoscopies
  ×100.
To assess and compare the costs associated with AI-assisted colonoscopy versus conventional colonoscopy. | During procedure (5minutes)
  Each cost associated with each examination, whether using AI-assisted or conventional colonoscopy, will be recorded prospectively.

CONTACTS AND LOCATIONS:
Overall Officials: Per Hedenstrom, MD. Ph D, Study Director — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Gothenbburg, Sweden

IPD SHARING:
Plan to Share IPD: No